CLINICAL TRIAL: NCT03607396
Title: Study for Evaluating the Real Use of Inhaled Aztreonam Lysine in Patients With Cystic Fibrosis
Acronym: REALIZA-FQ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: AFP-AZT-2017-01
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this observational trial is to evaluate the pulmonary function in cystic fibrosis patients that have been treated with inhaled aztreonam lysine comparing the previous 12 months before the treatment and the forward 12 months after initiating the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 6 years old that have been treated with Aztreonam Lysine (AZLI) at any time within 12 months before starting the treatment
* Diagnosis of Cystic Fibrosis confirmed
* Chronic infection by Pseudomonas aeruginosa
* Patients can be treated with any inhaled antibiotic before or after AZLI treatment
* Patients have to have the following FEV1 measures: 12 months before starting AZLI; at AZLI initiation; 12 months after starting AZLI
* For lung transplant patiens, only data before the transplant will be collected.

Exclusion Criteria:

* Non applicable

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cystic fibrosis patients colonized by Pseudomonas aeruginosa
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
FEV1 | 12 months
  Forced expiratory volume in one second (FEV1) measured during pulmonary function test.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Vall d'Hebron, Barcelona, Catalonia
  - Hospital La Fe, Valencia, Valencia
  - Hospital 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No